CLINICAL TRIAL: NCT04722861
Title: Development of the Glaucoma Visual Functioning Questionnaire-40 and Its Psychometric Properties
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020KYPJ186
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Primary Glaucoma; Glaucoma Suspect
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Glaucoma: Patients with primary glaucoma diagnosed by glaucoma professionals
  Interventions: Other: GVFQ-40
- Glaucoma Suspect Controls: Glaucoma suspect controls had a diagnosis of glaucoma suspect or ocular hypertension, and also were required to have a presenting Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity of 20/40 or better in both eyes.
  Interventions: Other: GVFQ-40

INTERVENTIONS:
Other: GVFQ-40 — GVFQ-40 is a 40-item questionnaire developed to evaluate the visual ability of glaucoma patients in detail. It consists of 40 items and measures the impact of glaucoma on restriction of participation in daily activities in five domains of functioning. Each item is rated on a five-level scale from ''no difficulty'' to ''can't do because of vision''. Another possible response is that the activity is not performed for nonvisual reasons.

SUMMARY:
The objective of this study is to develop and test the psychometric properties of a self-report questionaire, the Glaucoma Visual Functioning Questionnaire-40 (GVFQ-40), which was designed to measure the difficulty of daily activities of glaucoma patients and evaluate the effectiveness of clinical treatment or rehabilitation interventions.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness in the world. It is estimated that by 2040, the number of glaucoma patients in the world's population aged 40-80 will exceed 110 million [1]. As a chronic progressive blindness disease, glaucoma can seriously damage visual function such as visual acuity, visual field and contrast sensitivity, restrict patients' daily life activities and leads to a serious decline in vision-related quality of life (VRQOL) and health-related quality of life (HRQOL) [2-5]. Comprehensive evaluation of the visual function of glaucoma patients can not only educate the impact of glaucoma, but also reflect the effect of clinical treatment or rehabilitation interventions. However, the objective testing methods commonly used in clinic, such as visual acuity, visual field and contrast sensitivity, can only be used to evaluate part of the visual function of patients, which can not reflect the impact of disease and corresponding interventions from the point of view of patients. The use of patient defined measures of vision function in ophthalmic assessment and treatment evaluation is now well accepted and a number of questionnaires have been developed, such as NEI VFQ-25, LVQOL and SF-36, which mostly focus on investigating VRQOL or HRQOL[6-10]. There are comparatively few vision function questionnaires developed to measure the visual ability for glaucoma patients. The objective of this study is to develop and test the psychometric properties of a self-report questionaire, the Glaucoma Visual Functioning Questionnaire-40 (GVFQ-40), which was designed to measure the difficulty of daily activities of glaucoma patients and evaluate the effectiveness of clinical treatment or rehabilitation interventions.

The GVFQ-40 consists of 40 items and measures the impact of glaucoma on restriction of participation in daily activities in five domains of functioning (mobility, visual tracking, reading, identification and night vision ). Each item has six answer options, that is, no difficulty (score = 1), mild difficulty (score = 2), moderate difficulty (score = 3), extremely difficult (score = 4), completely unable to complete (score = 5), and do not performed for nonvisual reasons (no score).

ELIGIBILITY:
Inclusion Criteria:

1.1 Inclusion criteria of primary glaucoma group:

1. age ≥ 18 years old;
2. being able to express clearly and cooperate with the investigators;
3. diagnosed with primary glaucoma;
4. complete clinical data.

1.2 Inclusion criteria of glaucoma suspect controls:

1. age ≥ 18 years old;
2. being able to express clearly and cooperate with the investigators;
3. diagnosed with glaucoma suspect or ocular hypertension;
4. having a presenting Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity of 20/40 or better in both eyes;
5. complete clinical data.

Exclusion Criteria:

1.1 Exclusion criteria for primary glaucoma group:

1. serious cognitive dysfunction, psychological dysfunction, or hearing impairment;
2. physical motor dysfunction, hyperthyroidism or hypothyroidism, malignant tumors and other serious systemic diseases;
3. complicated with other ophthalmopathy affecting visual function (except cataract, ametropia), such as age-related macular degeneration, diabetic retinopathy, optic nerve disease, retinal vascular disease, etc;
4. surgical intervention (incisional or laser) within 2 weeks of the date of completing questionnaires (before or after);
5. not complete the questionnaire.

1.2 Exclusion criteria for glaucoma suspect controls:

1. serious cognitive dysfunction, psychological dysfunction, or hearing impairment;
2. physical motor dysfunction, hyperthyroidism or hypothyroidism, malignant tumors and other serious systemic diseases;
3. complicated with other ophthalmopathy affecting visual function (except cataract, ametropia), such as age-related macular degeneration, diabetic retinopathy, optic nerve disease, retinal vascular disease, etc;
4. not complete the questionnaire.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Primary glaucoma: patients with primary glaucoma diagnosed by glaucoma professionals
  2. Glaucoma Suspect Controls: glaucoma suspect controls had a diagnosis of glaucoma suspect or ocular hypertension, and also were required to have a presenting Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity of 20/40 or better in both eyes.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
GVFQ-40 | 1 day (Only once)
  GVFQ-40 is a 40-item questionnaire developed to evaluate the visual ability of glaucoma patients in detail. It consists of 40 items and measures the impact of glaucoma on restriction of participation in daily activities in five domains of functioning. Each item is rated on a five-level scale from ''no difficulty'' to ''can't do because of vision''. Another possible response is that the activity is not performed for nonvisual reasons. The GVFQ-40 is administered by a trained interviewer to all enrolled participants. A subset of participants (35 subjects) will complete the GVFQ-40 twice 2 to 3 weeks apart.

SECONDARY OUTCOMES:
Diagnosis and treatment information of ophthalmopathy | 1 day (Only once)
  The diagnosis and treatment information of ophthalmopathy, such as disease diagnosis name, time, history of drug treatment and history of operation, were obtained from the hospital electronic medical record system or outpatient medical record data.
NEI VFQ-25 | 1 day (Only once)
  The National Eye Institute-Visual Function Questionnaire-25 (NEI VFQ-25) is a valid and reliable VRQOL questionnaire designed for persons who have chronic eye diseases or low vision.
ETDRS visual acuity | 1 day (Only once)
  The information of ETDRS visual acuity was obtained from the hospital electronic medical record system or outpatient medical record data.
Intraocular pressure | 1 day (Only once)
  The information of intraocular pressure was obtained from the hospital electronic medical record system or outpatient medical record data.
Automatic perimetry report | 1 day (Only once)
  Automatic perimetry reports were obtained from the hospital electronic medical record system or outpatient medical record data.
Pelli-Robson contrast sensitivity | 1 day (Only once)
  Pelli-Robson contrast sensitivity test card was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones L, Garway-Heath DF, Azuara-Blanco A, Crabb DP; United Kingdom Glaucoma Treatment Study Investigators. Are Patient Self-Reported Outcome Measures Sensitive Enough to Be Used as End Points in Clinical Trials?: Evidence from the United Kingdom Glaucoma Treatment Study. Ophthalmology. 2019 May;126(5):682-689. doi: 10.1016/j.ophtha.2018.09.034. Epub 2018 Sep 28. PMID 30273622
- [Result] Sivaprasad S, Tschosik E, Kapre A, Varma R, Bressler NM, Kimel M, Dolan C, Silverman D. Reliability and Construct Validity of the NEI VFQ-25 in a Subset of Patients With Geographic Atrophy From the Phase 2 Mahalo Study. Am J Ophthalmol. 2018 Jun;190:1-8. doi: 10.1016/j.ajo.2018.03.006. Epub 2018 Mar 10. PMID 29530781
- [Derived] Huang H, Lin J, Luo M, Li Z, Zhu Y, Han J, Jin L, Li Y, Zhuo Y. Development and validation of the 40-item Glaucoma Visual Functioning Questionnaire. Br J Ophthalmol. 2023 Aug;107(8):1086-1091. doi: 10.1136/bjophthalmol-2021-320985. Epub 2022 Apr 4. PMID 35379597
- See also: VFQ-25 — https://pubmed.ncbi.nlm.nih.gov/29530781/
- See also: Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/30273622/